CLINICAL TRIAL: NCT05261854
Title: Effects of Pressure Biofeedback on Deep Cervical Flexor Muscle Training for Neck Pain, Functional Disability and Muscle Endurance Among University Teachers. A Randomized Control Trail
Brief Title: Effect Of Pressure Biofeedback on Deep Cervical Muscle Training Among University Teachers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC-FSD-00246
Record Dates: First submitted 2022-02-20; First posted 2022-03-02 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Neck Pain
Keywords: Neck pain; Disabilty; Muscle endurance; Pressure biofeedback; Teachers
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The study Would be double blind as the identity of patients group will not be revealed to the assessor and the patient will also be unaware of group to which they will be allocated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep cervical muscle training using pressure biofeedback and conventional Exercises (Experimental): The duration of preesure biofeedback includes 3 sets in a session with 10 repetitions each with 2 minutes of rest between sets and 5 days a week for 6 weeks.
  Conventional exercises like Stretching and strengthening of neck flexor muscles will include 10 repetitions, each held for 10s with rest of 2 minutes between sets. The session will be conducted for 6 weeks, 5 days a week.
  Interventions: Device: Pressure biofeedback
- conventional exercises for Neck pain (Experimental): Only conventional exercises like stretching and strengthening of neck flexor muscles will be given.
  Interventions: Other: Conventional exercises for deep cervical muscle training

INTERVENTIONS:
Device: Pressure biofeedback — Deep cervical flexor training by using preesure biofeedback will be given 5 days a week for 6 week Conventional exercise for deep cervical muscle training will be given 5 days a week for 6 weeks
  Arms: Deep cervical muscle training using pressure biofeedback and conventional Exercises
Other: Conventional exercises for deep cervical muscle training — Conventional exercise for deep cervical muscle training will be given 4 days a week for 6 weeks
  Arms: conventional exercises for Neck pain

SUMMARY:
The aim of this study is to investigate the effect of pressure biofeedback on deep cervical muscle in university teachers suffering from neck pain, Functional Disability and muscle endurance.

DETAILED DESCRIPTION:
The purpose of this study will be to determine whether training of deep cervical flexor muscles with pressure biofeedback has any significant advantage over conventional training for pain and disability experienced by university teachers with neck pain. This study will be a randomized control trial with double blinded protocol. Patient will be randomly allocated in two groups. the experimental group received deep cervical flexor muscles training with pressure biofeedback and conventional exercises. The control group received deep cervical flexor muscles training with only conventional exercises.

ELIGIBILITY:
Inclusion Criteria:

* Both gender
* age between 24 to 45 years
* At least 4 years of teaching experience and average 8 hours of working per day
* Chronic Neck pain score of more than 5 on numeric pain rating scale
* Mild to moderate disability Score on neck disability index

Exclusion Criteria:

* Participants with any ongoing treatment for neck pain
* History of cervical spine surgery or reported any neurological signs.
* History of any congenital or acquired postural deformity, spinal cord compression, tumour, instability, fracture, inflammatory disease or infection.

Ages: 24 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-04-05 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating Scale | 8th week
  Numeric pain rating scale used to determine pain intensity experienced by individuals. It consist of a horizontal or vertical line with total of 11 numbers,ranging from 0 to 10. Where 0 indicates no pain while 10 is the worst pain.
Inclinometer | 8th week
  It is an instrument used for measuring the angles of tilt,elevation and depression of an object with respect to gravity.
Cranio-cervical flexion test | 8th week
  It is a clinical test of the anatomical action of the deep cervical flexor muscles. It could be described as a test of neuromotor control. The features assessed are the activation and isometric endurance of the deep cervical flexors
Neck Disability index | 8th week
  This questionnaire has been designed to give us information as to how your neck pain has affected your ability to manage in everyday life.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Riphah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No